CLINICAL TRIAL: NCT05506995
Title: Tissue-resident Memory T Cells Expression Among the Repigmentation Patterns Induced by NB-UVB Phototherapy in Vitiligo
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Clinical and research professor in Dermatology, Universidad Autonoma de San Luis Potosí
Other Study IDs: 63-21
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Vitiligo
Keywords: vitiligo; Ultraviolet Therapy; Pigmentation; Tissue-resident memory T cells; Hobbit; Blimp1; Runx3; Notch1
MeSH Terms: conditions — Vitiligo; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Vitiligo vulgaris: A serial of vitiligo patients under treatment with UVB-NB

SUMMARY:
Vitiligo is the most commonly acquired depigmentation disorder characterized by selective destruction of melanocytes resulting in well-circumscribed achromic macules. Tissue-resident memory T cells (TRM) are memory T lymphocyte subsets that reside in the skin, lack recirculation, proliferate locally, produce cytokines, and may be implicated in relapses. NB-UVB Phototherapy induces repigmentation in certain patterns. The aim of this study was to determine the levels of TRM cells on vitiligo lesions, and after phototherapy by repigmentation pattern.

DETAILED DESCRIPTION:
Vitiligo is the most commonly acquired depigmentation disorder characterized by the selective destruction of melanocytes. Its etiology is not yet fully understood, but the most accepted hypotheses are genetic predisposition, environmental factors, oxidative stress and immune response. In relation with the latter, the damage-associated molecular patterns activate TRM cells and induce interferon-gamma that release CXCL9/10, recruiting cytotoxic CD8+ that ultimately destroys melanocytes. Furthermore, the lesions recur 40% in the first year and in the same site, suggesting local autoimmune response by TRM cells.

The TRM cells are memory T lymphocyte subsets that reside in the skin, lack recirculation, proliferate locally, and produce cytokines. TRM cells express the CD69+CD103+ surface markers. Moreover, TRM cells express specific transcription factors like Hobbit, Blimp1, Runx3 and Notch1, which regulate their differentiation and survival.

Interleukin (IL)-15 stimulates Hobbit, which drives TRM cells long-term maintenance by blocking CCR7-S1PR1 and promoting the expression of CD103+. Blimp1 is essential for the differentiation of TRM cells, as it inhibits the differentiation of naive T cells into circulating-memory T cells, and regulates the effector function by stimulating granzyme B and promoting the expression of CD69+. Runx3 is essential for TRM cells long-term maintenance by promoting CD103+, which can also induce Blimp1 and Hobbit. Notch1 is essential for the maintenance of CD103+, facilitating the TRM-epithelium linking. Both TRM cells and central-memory T cells have been found in vitiligo lesions, and the CD69+CD103+ TRM cells are increased in vitiligo skin.

NB-UVB phototherapy is the first line treatment for vitiligo involving more than 10 percent of the body surface area, with an average response rate of 67%. It promotes repigmentation by differentiation and migration of perilesional melanocytes, tyrosinase increase and inhibition of effector and memory T cells. NB-UVB promotes different patterns of repigmentation such as follicular, marginal, and diffuse. The NB-UVB exposure causes a decrease in the transforming factor beta that maintain the expression of CD103+, but there is no data about the CD69+ modification, suggesting a possible effect on TRM cells.

Vitiligo relapses tend to be at the same site of previous lesions, suggesting local autoimmunity by the TRM cells that could be modified by UVB-NB phototherapy. Phototherapy can inhibit effector and memory-T cells; however its effect on TRM cells in vitiligo and their modification is unknown. The purpose of this study was to determine the levels of TRM cells on vitiligo lesions, and following NB-UVB phototherapy by repigmentation pattern.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Symmetric vitiligo
* Affected body surface greater than 10%
* Patients with follicular, marginal and diffuse repigmenting patterns
* No previous topical or systemic treatment in the previous 2 and 3 months, respectively
* Signed informed consent

Exclusion Criteria:

* Concomitant treatment or systemic diseases
* Pregnancy
* Drugs intake
* Mental disorders
* Acral, universal or segmental vitiligo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis of vitiligo vulgaris with more than 10 percent of the total body surface affected.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Tissue-resident memory T cells | Up to 1 year
  To quantify the expression of Tissue-resident memory T cells before and after phototherapy

SECONDARY OUTCOMES:
Tissue-resident memory T cells among the repigmentation patterns | Up to 1 year
  To quantify the expression of Tissue-resident memory T cells among the repigmentation patterns induced by NB-UVB phototherapy
Arrangment of the Tissue-resident memory T cells among the repigmentation patterns | Up to 1 year
  To show and quantify the fluorescence intensity of the CD69+CD103+ TRM cells among the repigmentation patterns induced by NB-UVB phototherapy
TRM transcriptional factors profile | Up to 1 year
  To quantify the TRM transcriptional factors expression in lesional skin and between the repigmentation patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Castanedo-Cazares, MD, Principal Investigator — Universidad Autonoma de San Luis Potosi
Locations (1):
- Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bae JM, Jung HM, Hong BY, Lee JH, Choi WJ, Lee JH, Kim GM. Phototherapy for Vitiligo: A Systematic Review and Meta-analysis. JAMA Dermatol. 2017 Jul 1;153(7):666-674. doi: 10.1001/jamadermatol.2017.0002. PMID 28355423
- [Result] Fraczek A, Owczarczyk-Saczonek A, Placek W. The Role of TRM Cells in the Pathogenesis of Vitiligo-A Review of the Current State-Of-The-Art. Int J Mol Sci. 2020 May 18;21(10):3552. doi: 10.3390/ijms21103552. PMID 32443482
- [Result] Riding RL, Harris JE. The Role of Memory CD8+ T Cells in Vitiligo. J Immunol. 2019 Jul 1;203(1):11-19. doi: 10.4049/jimmunol.1900027. PMID 31209143
- [Result] Richmond JM, Strassner JP, Rashighi M, Agarwal P, Garg M, Essien KI, Pell LS, Harris JE. Resident Memory and Recirculating Memory T Cells Cooperate to Maintain Disease in a Mouse Model of Vitiligo. J Invest Dermatol. 2019 Apr;139(4):769-778. doi: 10.1016/j.jid.2018.10.032. Epub 2018 Nov 10. PMID 30423329
- [Result] Behr FM, Chuwonpad A, Stark R, van Gisbergen KPJM. Armed and Ready: Transcriptional Regulation of Tissue-Resident Memory CD8 T Cells. Front Immunol. 2018 Jul 30;9:1770. doi: 10.3389/fimmu.2018.01770. eCollection 2018. PMID 30131803
- [Result] Mackay LK, Minnich M, Kragten NA, Liao Y, Nota B, Seillet C, Zaid A, Man K, Preston S, Freestone D, Braun A, Wynne-Jones E, Behr FM, Stark R, Pellicci DG, Godfrey DI, Belz GT, Pellegrini M, Gebhardt T, Busslinger M, Shi W, Carbone FR, van Lier RA, Kallies A, van Gisbergen KP. Hobit and Blimp1 instruct a universal transcriptional program of tissue residency in lymphocytes. Science. 2016 Apr 22;352(6284):459-63. doi: 10.1126/science.aad2035. PMID 27102484
- [Result] Zubair R, Hamzavi IH. Phototherapy for Vitiligo. Dermatol Clin. 2020 Jan;38(1):55-62. doi: 10.1016/j.det.2019.08.005. Epub 2019 Oct 18. PMID 31753192
- [Result] Castanedo-Cazares JP, Cortes-Garcia JD, Fuentes-Ahumada C, Martinez-Rosales K, Torres-Alvarez B. Repigmentation patterns induced by NB-UVB and their relationship with melanocytic migration and proliferation in vitiligo. Photodermatol Photoimmunol Photomed. 2016 Sep;32(5-6):269-275. doi: 10.1111/phpp.12275. Epub 2016 Oct 5. PMID 27627998
- [Result] Patra V, Laoubi L, Nicolas JF, Vocanson M, Wolf P. A Perspective on the Interplay of Ultraviolet-Radiation, Skin Microbiome and Skin Resident Memory TCRalphabeta+ Cells. Front Med (Lausanne). 2018 May 30;5:166. doi: 10.3389/fmed.2018.00166. eCollection 2018. PMID 29900173
- [Result] Azzolino V, Zapata L Jr, Garg M, Gjoni M, Riding RL, Strassner JP, Richmond JM, Harris JE. Jak Inhibitors Reverse Vitiligo in Mice but Do Not Deplete Skin Resident Memory T Cells. J Invest Dermatol. 2021 Jan;141(1):182-184.e1. doi: 10.1016/j.jid.2020.04.027. Epub 2020 May 25. No abstract available. PMID 32464150